CLINICAL TRIAL: NCT01682213
Title: A Phase 2 Trial of Adjuvant Dabrafenib (GSK2118436) in Patients With Surgically Resected AJCC Stage IIIC Melanoma Characterized by a BRAFV600E/K Mutation
Brief Title: Adjuvant Dabrafenib (GSK2118436) in Patients With Surgically Resected AJCC Stage IIIC Melanoma Characterized by a BRAFV600E/K Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-124
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
Keywords: Dabrafenib; (GSK2118436); BRAFV600E/K; Resected AJCC Stage IIIC; 12-124
MeSH Terms: conditions — Melanoma | interventions — dabrafenib

ARMS (1):
- dabrafenib (Experimental): This is a single institution phase II trial assessing the efficacy of adjuvant dabrafenib (GSK2118436) in patients with surgically resected AJCC stage IIIC melanoma characterized by a BRAFV600E/K mutation.
  Interventions: Drug: Dabrafenib

INTERVENTIONS:
Drug: Dabrafenib — Following definitive surgical resection, eligible patients will receive dabrafenib at 150 mg twice a day by mouth for 4 cycles (± 5 days). One cycle is 28 days.

SUMMARY:
In this study, the investigator's want to find out if dabrafenib can stop stage IIIC melanoma from coming back after surgery.

ELIGIBILITY:
Inclusion Criteria:

* AJCC (2009) stage IIIC cutaneous melanoma rendered free of disease by surgical resection no greater than 90 days prior study enrollment. Patients with unknown primaries will be eligible for this trial. Patients with a history of resected stage I or II cutaneous melanoma who subsequently have their first disease recurrence meeting the criteria for stage IIIC disease will also be eligible for this trial.
* Patients must have clear margins after wide local excision. Patients with nodes that are palpable or detectable on radiologic imaging must have an adequate lymphadenectomy.
* Patients must be adequately recovered from surgery, radiation therapy, or any surgical complications prior to enrollment. In general, this means patients will be off antibiotics from wound infections and drains removed. However, if necessary, patients can be treated with a drain in place at the discretion of the PI if the 90 days window is about to expire.
* Histologic proof of melanoma reviewed and confirmed by MSKCC.
* A documented BRAFV600E or BRAFV600K mutation by genotyping or IHC [35]performed by a CLIA certified laboratory.
* Age ≥ 16 years old
* ECOG performance status = 0 or Karnofsky Performance Status equivalent
* The ability to swallow pills.
* Patients must have adequate organ and marrow function as defined below:

Absolute neutrophil count ≥1.5 K/mcL Platelets ≥ 100 K/mcL Hemoglobin ≥ 9.0 g/dL Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)

≤ 3.0 X institutional ULN if the patient has Gilbert's Syndrome AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN Creatinine ≤ 1.5 X institutional ULN or creatinine clearance (calculated or measured) > 60 ml/min

* Women with child bearing potential and men with reproductive potential must be willing to practice acceptable methods of contraception.

Exclusion Criteria:

* Patients with a history of stage III melanoma (any primary melanoma with locoregional nodal/subcutaneous disease) treated with surgical resection who subsequently have disease recurrence meeting the criteria for stage IIIC disease.
* Prior therapy with ipilimumab, other BRAF inhibitors, or MEK inhibitors.
* Concurrent adjuvant immunotherapy, chemotherapy, or radiotherapy.
* Current use of a prohibited medication while on dabrafenib
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs.
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Pregnant women and lactating women.
* A concurrent second malignancy even if it does not require active therapy. Patients with indolent B-cell malignancies will not be eligible. Prior malignancy will be allowed as long as the patient is known to be free of disease for at least 3 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* QTc interval > 500 msec unless a bundle branch block is also present.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dabrafenib
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dabrafenib
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 54 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse Free Survival
Description: Relapse free survival is defined as the time from surgical resection to the first recurrence or death as assessed by physical examination and radiographic evaluation. All recurrences will be confirmed by biopsy and histologic evaluation.
Time Frame: 24 months
Population: 2 participants withdrew consent 1 week after signing consent
Measure: Number; unit: percentage of participants
Arm/Group | Dabrafenib
Number analyzed (Participants) | 21
percentage of participants | 28.6

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from surgical resection to death or last follow-up.
Time Frame: 2 years
Population: 2 participants withdrew consent 1 week after signing consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dabrafenib
Number analyzed (Participants) | 21
percentage of participants | 78 [51 to 91]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity will be graded by the NCI Common Toxicity Criteria (CTC) version 4.0 with each cycle of adjuvant dabrafenib.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dabrafenib
All-Cause Mortality (participants affected / at risk) | 8/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib (N=23)
Anemia (Blood and lymphatic system disorders) | 1
Chills (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 2
Neoplasms ben/mal/unk (inccyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Platelet count decreased (Investigations) | 1
Seizure (Nervous system disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib (N=23)
Rash (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 7
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Flushing (Vascular disorders) | 3
New primary melanoma (Skin and subcutaneous tissue disorders) | 1
Abducens nerve disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 2
Photophobia (Eye disorders) | 1
Blurred vision (Eye disorders) | 2
Headache (Nervous system disorders) | 8
Diarrhea (Gastrointestinal disorders) | 4
Nausea/Vomiting (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Leukopenia (Investigations) | 5
Transaminitis (Investigations) | 1
Fatigue (General disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 7
Insomnia (Psychiatric disorders) | 1
Chills (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT01682213/Prot_SAP_000.pdf